CLINICAL TRIAL: NCT00961831
Title: Open-label, Multicenter Study for an Evaluation of Radiation Dosimetry, Metabolism, Safety and Tolerability of the [F18] Labeled PET (Positron Emission Tomography) Tracer BAY 85-8050 Following a Single Intravenous Administration in Healthy Volunteers, as Well as the Investigation of Safety, Tolerability and Diagnostic Performance of the Tracer in PET/CT (Computer Tomography) in Patients
Brief Title: Radiation Dosimetry, Metabolism, Safety, Tolerability and Positron Emission Tomography/Computed Tomography (PET/CT) Imaging With BAY 85-8050 in Healthy Volunteers and Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13107; 2008-000962-21 (EudraCT Number)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Neoplasm
Keywords: Neoplasm; PET/CT diagnosis; PET tracer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: F-18 (BAY85-8050)
- Arm 2 (Experimental)
  Interventions: Drug: F-18 (BAY85-8050)

INTERVENTIONS:
Drug: F-18 (BAY85-8050) — Cancer patients, injection of BAY 85-8050, PET/CT
  Arms: Arm 1
Drug: F-18 (BAY85-8050) — Healthy volunteers, injection of BAY 85-8050, whole body PET/CT for determination of effective dose, kinetics of BAY 85-8050 in blood
  Arms: Arm 2

SUMMARY:
This study is a visual assessment of diagnostic PET/CT images obtained after a single intravenous injection of BAY85-8050 in patients with cancer

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers only
* Males/females, >/=50 and </= 65 years of age
* Cancer patients only
* Males/females >/= 35 years and </= 75 years of age
* Patient had an FDG PET/CT for detection, or staging, or restaging, or therapy response assessment that still showed tumor mass

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable other medical disease (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY85-8050, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
* Known sensitivity to the study drug or components of the preparation

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2009-12-16 (Actual); Study Completion 2009-12-16 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesions | Within up to 2 hours after treatment

SECONDARY OUTCOMES:
Quantitative analysis of BAY 85-8050 uptake into lesions (Standardized Uptake Values, SUVs) | Within up to 2 hours after treatment
Serum chemistry:Glutamate pyruvate transaminase (GPT/ALAT), gamma-glutamyl transferase (gamma-GT), glutamate-oxaloacetate transaminase (GOT), alkaline phosphatase, total bilirubin, creatinine, total protein | At least 2 times within 8 days after treatment
Electrocardiogram (ECG) | at least 2 times within 8 days after treatment
Vital signs: Heart rate, blood pressure | at least 2 times within 8 days after treatment
Adverse events collection | continuously for at least 8 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- München, Bavaria, Germany